CLINICAL TRIAL: NCT00969098
Title: Early Response Evaluation in Malignant Pleural Mesothelioma By Total Glycolytic Volume (TGV) Analysis of Serial FDG-PET Scans (Positron Emission Tomography Scans)
Brief Title: Response Evaluation in Malignant Pleural Mesothelioma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: ONC/OSS-02/2009
Record Dates: First submitted 2009-08-06; First posted 2009-08-31 (Estimated); Last update posted 2015-08-06 (Estimated); Status verified 2015-08

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Histologically proven of Malignant pleural mesothelioma;; Patients not candidate to radical surgery;; Candidate to first-line pemetrexed-based chemotherapy;
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Recently, a few small trials have shown promising results on value of fluoro-2-deoxy-D-glucose and positron emission tomography imaging in response assessment in Malignant Pleural Mesothelioma. These studies considered different parameters in Positron Emission Tomography (PET) analysis, mainly the standardized uptake value and volume-based parameters such as total glycolytic volume.

DETAILED DESCRIPTION:
This is a retrospective analysis of two consecutive and homogeneous series of Malignant Pleural Mesothelioma patients treated with first-line pemetrexed-based chemotherapy and evaluated by CT scan and FDG-PET.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven MALIGNANT PLEURAL MESOTHELIOMA
* Patients not candidate to radical surgery
* Unidimensionally and/or bidimensionally CT-measurable disease and Candidate to first-line pemetrexed-based chemotherapy

Exclusion Criteria:

* Histologically not proven MALIGNANT PLEURAL MESOTHELIOMA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically proven MALIGNANT PLEURAL MESOTHELIOMA and Patients not candidate to radical surgery
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-06; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
To validate a semi-automated iterative threshold-based region growing algorithm in a previously published series of patients. | 4 months

SECONDARY OUTCOMES:
To extend the analysis to another series of consecutive patients with MALIGNANT PLEURAL MESOTHELIOMA treated with first-line pemetrexed-based chemotherapy, and to perform a combined analysis of the two groups. | 4 months
To validate the new liver-based threshold semi-automated algorithm on the GE ADW4.6 workstation with the algorithm validated in step 1 in the same subset of patients. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Background] Robinson BW, Musk AW, Lake RA. Malignant mesothelioma. Lancet. 2005 Jul 30-Aug 5;366(9483):397-408. doi: 10.1016/S0140-6736(05)67025-0. PMID 16054941
- [Background] Sugarbaker DJ, Flores RM, Jaklitsch MT, Richards WG, Strauss GM, Corson JM, DeCamp MM Jr, Swanson SJ, Bueno R, Lukanich JM, Baldini EH, Mentzer SJ. Resection margins, extrapleural nodal status, and cell type determine postoperative long-term survival in trimodality therapy of malignant pleural mesothelioma: results in 183 patients. J Thorac Cardiovasc Surg. 1999 Jan;117(1):54-63; discussion 63-5. doi: 10.1016/s0022-5223(99)70469-1. PMID 9869758
- [Background] Vogelzang NJ, Rusthoven JJ, Symanowski J, Denham C, Kaukel E, Ruffie P, Gatzemeier U, Boyer M, Emri S, Manegold C, Niyikiza C, Paoletti P. Phase III study of pemetrexed in combination with cisplatin versus cisplatin alone in patients with malignant pleural mesothelioma. J Clin Oncol. 2003 Jul 15;21(14):2636-44. doi: 10.1200/JCO.2003.11.136. PMID 12860938
- [Background] Ceresoli GL, Zucali PA, Favaretto AG, Grossi F, Bidoli P, Del Conte G, Ceribelli A, Bearz A, Morenghi E, Cavina R, Marangolo M, Parra HJ, Santoro A. Phase II study of pemetrexed plus carboplatin in malignant pleural mesothelioma. J Clin Oncol. 2006 Mar 20;24(9):1443-8. doi: 10.1200/JCO.2005.04.3190. PMID 16549838
- [Background] Ceresoli GL, Chiti A, Zucali PA, Cappuzzo F, De Vincenzo F, Cavina R, Rodari M, Poretti D, Lutman FR, Santoro A. Assessment of tumor response in malignant pleural mesothelioma. Cancer Treat Rev. 2007 Oct;33(6):533-41. doi: 10.1016/j.ctrv.2007.07.012. Epub 2007 Aug 30. PMID 17764849
- [Background] Byrne MJ, Nowak AK. Modified RECIST criteria for assessment of response in malignant pleural mesothelioma. Ann Oncol. 2004 Feb;15(2):257-60. doi: 10.1093/annonc/mdh059. PMID 14760119
- [Background] Flores RM, Akhurst T, Gonen M, Zakowski M, Dycoco J, Larson SM, Rusch VW. Positron emission tomography predicts survival in malignant pleural mesothelioma. J Thorac Cardiovasc Surg. 2006 Oct;132(4):763-8. doi: 10.1016/j.jtcvs.2006.03.068. PMID 17000285
- [Background] Flores RM, Akhurst T, Gonen M, Larson SM, Rusch VW. Positron emission tomography defines metastatic disease but not locoregional disease in patients with malignant pleural mesothelioma. J Thorac Cardiovasc Surg. 2003 Jul;126(1):11-6. doi: 10.1016/s0022-5223(03)00207-1. PMID 12878934
- [Background] Weber WA. Use of PET for monitoring cancer therapy and for predicting outcome. J Nucl Med. 2005 Jun;46(6):983-95. PMID 15937310
- [Background] Ceresoli GL, Chiti A, Zucali PA, Rodari M, Lutman RF, Salamina S, Incarbone M, Alloisio M, Santoro A. Early response evaluation in malignant pleural mesothelioma by positron emission tomography with [18F]fluorodeoxyglucose. J Clin Oncol. 2006 Oct 1;24(28):4587-93. doi: 10.1200/JCO.2006.06.8999. PMID 17008700